CLINICAL TRIAL: NCT06805331
Title: The Effect of Health Belief Model-Based Pelvic Floor Muscle Exercise Training on Urinary Incontinence and Quality of Life in Female Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nurgül KAPLAN (Other)
Responsible Party: Sponsor-Investigator, Nurgül KAPLAN, Instructor, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GaziosmanpasaU- HMŞRLK-NK-01
Record Dates: First submitted 2025-01-09; First posted 2025-02-03 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis; Urinary Incontinence
Keywords: Exercise training; Multiple Sclerosis; Pelvic Floor Muscle Exercise; Health Belief Model; Urinary Incontinence; Quality of Life
MeSH Terms: conditions — Multiple Sclerosis; Urinary Incontinence | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized-controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which group they are in. The person who analyzes the data obtained at the end of the study will not know the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Pelvic Floor Muscle Exercise Training) (Experimental): The researcher will explain pelvic floor muscle exercises to the patients within the framework of the health belief model. After the pelvic floor muscle exercise training is given, the patients will be asked to do these exercises three times a day (morning-afternoon-evening) for three months (12 weeks).
  Interventions: Behavioral: Intervention group(Pelvic Floor Muscle Exercise Training)
- No Intervention (Control Group) (Other): Participants in the control group will undergo standard care procedures without receiving any intervention. The results will be evaluated for comparison purposes.
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: Intervention group(Pelvic Floor Muscle Exercise Training) — The intervention will involve educating participants on pelvic floor muscle exercises, using the health belief model. The goal is to evaluate improvements in incontinence severity, quality of life, and pelvic floor muscle exercise self-efficacy
  Arms: Intervention Group (Pelvic Floor Muscle Exercise Training)
Other: control group — Participants in the control group will continue to receive their current standard of care and will not receive any additional interventions.
  Arms: No Intervention (Control Group)

SUMMARY:
The aim of this study is to evaluate the effect of Pelvic Floor Muscle Exercise Training According to the Health Belief Model on Urinary Incontinence and Quality of Life in Female Patients with Multiple Sclerosis.

Hypothesis 01: Pelvic floor muscle exercise training applied using the health belief model is not effective in reducing urinary complaints in female MS patients.

Hypothesis 1: Pelvic floor muscle exercise training applied using the health belief model is effective in reducing urinary complaints in female MS patients.

Hypothesis 02: Pelvic floor muscle exercise training applied using the health belief model is not effective on the quality of life of female MS patients.

Hypothesis 2: Pelvic floor muscle exercise training applied using the health belief model is effective on the quality of life of female MS patients.

DETAILED DESCRIPTION:
This study will be conducted to evaluate the effect of pelvic floor muscle exercise (PFMT) training on urinary incontinence and quality of life in women with multiple sclerosis (MS) according to the health belief model (HBM). This study will be conducted as a randomized controlled experimental study with 46 women with urinary incontinence complaints who were diagnosed with MS and followed up at the MS outpatient clinic of the Neurology Department of Tokat Gaziosmanpaşa University Hospital. Patients will be included in the control (23) and intervention (23) groups by simple randomization method. In collecting the research data; Questionnaire on Descriptive Characteristics, International Incontinence Questionnaire Short Form (ICIQ-SF), Incontinence Quality of Life Scale (I-QOL), Incontinence Severity Index (ISI), Broome Pelvic Floor Muscle Exercise Self-Efficacy Scale (Broome PMSES), Expanded Disability Status Scale (EDSS), Bladder diary will be used. The research data will be collected after the experimental and control groups are determined after the approval. Data collection forms will be applied to both groups at the beginning of the study and at the end of the 1st and 3rd months. Patients in the intervention group will perform pelvic floor muscle exercises 3 times a day (morning-afternoon-evening) for 3 months. No intervention will be applied to patients in the control group. The data will be entered into a statistical package program and evaluated. No study has been found in the literature evaluating the effect of PTCE training according to the SIM on urinary incontinence and quality of life in female patients with MS. The research has original value in this respect and will contribute scientifically to national and international literature. If the research is successful, it is thought that PTCE training according to the health belief model in female patients with MS will be proven as a non-pharmacological intervention and will provide a new nursing intervention in the field. PTCE training according to the SIM in female patients with MS will reduce urinary incontinence and increase quality of life. In addition, it is thought that it will contribute positively to the physiological, psychological and social recovery process of MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old and above,
* Being a woman,
* Being diagnosed with MS,
* Having urinary incontinence,
* Not having an attack in the last thirty days,
* No change in medical treatment in the last three months,
* Being under 6.5 on the Expanded Disability Status Scale (EDSS),
* Not having a diagnosis of cognitive or mental disorder,
* Being willing to participate in the study,

Exclusion Criteria:

* Presence of pregnancy,
* Presence of urinary tract infection,
* Presence of another neurological disease that may cause incontinence,
* History of cancer,
* History of pelvic surgery,
* Presence of pelvic organ prolapse,
* Deficiency in evaluation parameters,
* Non-compliance with treatment programs,
* Change in drug treatment during treatment,
* Receiving PTCE in the last six months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — * Being a woman,
  * Being diagnosed with MS,
  * Having urinary incontinence,
Enrollment: 46 (Actual)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Urinary Incontinence | Three months
  Urinary incontinence severity and impact will be assessed at baseline and after 3 months using the International Incontinence Questionnaire Short Form (ICIQ-SF).

SECONDARY OUTCOMES:
Quality of life in Women with Multiple Sclerosis | Three months
  The impact of incontinence on quality of life will be assessed at baseline and after 3 months using the Incontinence Quality of Life Scale (I-QOL).

OTHER OUTCOMES:
The Broome Pelvic Floor Muscle Exercise Self-Efficacy | Three months
  Individuals' self-efficacy beliefs regarding performing pelvic floor muscle exercises will be assessed using the Broome Pelvic Floor Muscle Exercise Self-Efficacy Scale at baseline and after 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR